CLINICAL TRIAL: NCT00321113
Title: An Open, Multicentre, Randomised, Parallel Group Study to Compare in Marginal Old-for-old Renal Transplant Patients the Safety and Efficacy of Two Treatments: Sequential Mycophenolate Mofetil/Delayed Tacrolimus Plus Steroids vs Tacrolimus Plus Mycophenolate Mofetil in Patients Requiring Induction With Anti-IL2 Antibody
Brief Title: Comparison of Two Tacrolimus Based Immunosuppressive Regimens in Recipients Receiving Marginal Donor Kidneys
Acronym: TIGRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-02-IT-01
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: KIDNEY TRANSPLANTATION
Keywords: MARGINAL KIDNEY; TACROLIMUS; IMMUNOSUPPRESSION; ELDERLY RECEPIENTS
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): oral
  Interventions: Drug: tacrolimus; Drug: mycophenolate mofetil
- 2 (Experimental): oral
  Interventions: Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: steroids

INTERVENTIONS:
Drug: tacrolimus — immunosuppression
  Other Names: Prograf; FK506
Drug: mycophenolate mofetil — oral
  Other Names: MMF
Drug: steroids — oral
  Arms: 2

SUMMARY:
The purpose of this study is to explore the safety and efficacy of two different immunosuppressive regimens (sequential tacrolimus/mycophenolate mofetil [MMF] plus steroids versus tacrolimus plus MMF, following induction with daclizumab) in recipients of marginal donor kidneys.

DETAILED DESCRIPTION:
An open, multicentre, randomized, parallel group study to compare in marginal old-for-old renal transplant patients the safety and efficacy of two treatments: sequential mycophenolate mofetil/delayed tacrolimus plus steroids vs tacrolimus plus mycophenolate mofetil, in patients requiring induction with anti-IL2 monoclonal antibody.

Elderly (≥50 years) low risk patients (PRA grade ≤50%, in the previous 6 months) receiving an allograft transplantation of marginal kidney(s) from elderly (>65 years) donors (old-for-old allocation) will be randomized to one of the following treatment arms:

Arm1: Sequential mycophenolate mofetil/tacrolimus/steroids

Arm2: Tacrolimus/mycophenolate mofetil/steroid one single dose (perioperatively)

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients minimum 60 years of age undergoing a cadaveric kidney transplant
* Patient has end stage kidney disease and is a suitable candidate for primary renal transplantation.
* Donors older than 60 years
* Female patients of child bearing age agree to practice effective birth control during the study.
* Patient has been fully informed and has given written informed consent

Exclusion Criteria:

* Patient has significant, uncontrolled, concomitant infections and/or severe diarrhoea, vomiting, or active peptic ulcer
* Patient has previously received or is receiving an organ transplant other than kidney or a kidney retransplant
* Any pathology or medical condition that can interfere with this protocol study proposal
* Other exclusion criteria apply

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2004-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Calculated creatinine clearance | 6 months

SECONDARY OUTCOMES:
Acute Rejection, patient survival, graft survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (12):
- Italy (12):
  - Bologna
  - Cagliari
  - Milan
  - Modena
  - Padua
  - Palermo
  - Roma
  - Sassari
  - Siena
  - Treviso
  - Udine
  - Vicenza

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=199